CLINICAL TRIAL: NCT01025531
Title: Cell Bound Complement Activation Proteins as Markers of Liver Injury
Status: Withdrawn | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO08060224; physician funding (Other: UPMC)
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All biologic samples will be under the control of the principal investigator . To protect confidentiality, all personal identifiers will be removed and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with newly diagnosed Hepatitis C: Hepatitis C patients newly diagnosed

SUMMARY:
Subjects who eventually undergo treatment for HCV, we will gather treatment data (start and stop dates), and repeat CB-CAP analysis at weeks 4, 12, 24 and 72 (+/- 2 week window allowed at each time point) to determine whether CB-CAPs levels predict virologic response in treated subjects. Routine laboratory data will also be collected at these time points.

DETAILED DESCRIPTION:
The investigators will recruit consecutive HCV infected subjects from the Center for Liver Diseases (CLD) at the University of Pittsburgh Medical Center (UPMC) who are scheduled to undergo a liver biopsy as part of their routine clinical care. The liver biopsies will be read concurrently by a single study pathologist who is blinded to the subjects' clinical status. At the time of liver biopsy, blood will be drawn to perform CB-CAP assays. The CB-CAP levels will be correlated with the liver biopsy result to assess their ability to predict degree of liver injury. The investigators will retrieve labs done for routine clinical care closest to the time of liver biopsy, including complete blood count, serum aminotransferase levels, and a biochemical profile.

A total of 250 subjects will be recruited for this study. Data gathered would include demographic and clinical information, risk factors for HCV, information about drug and alcohol use and anthropometric measurements (height, weight, abdominal circumference, etc.).

For the subset of subjects who are then initiated on treatment for HCV by their healthcare providers, we will gather treatment information (start date, stop date, treatment regimen and dosage, etc.) and blood will be drawn at treatment weeks 4, 12, 24 and 72 (+/- 2 week window allowed at each time point) to determine whether CB-CAPs levels predict virologic response in treated subjects. Routine laboratory data will also be collected at these time points. The +/- 2 week time window is allowed so that the blood draw can be done at a routine clinical visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older at time of evaluation
* Able to give informed consent
* Confirmed HCV infection by standard antibody testing any time prior to enrollment
* Detectable HCV RNA in routine clinical testing any time prior to enrolment (since our aim is to determine the correlation between CB-CAPs and histologic activity in chronic HCV)
* Undergoing liver biopsy as part of their routine clinical care

Exclusion Criteria:

Any previous treatment for HCV

* Any other chronic or active liver disease that, in the opinion of the investigator, can affect liver histology (history of alcohol use in itself will not be an exclusion criteria)
* HIV coinfection
* Chronic Hepatitis B infection (HBsAg+ or HBeAg+ or HBV DNA+ upon last testing)
* Acute Hepatitis A infection (HAV IgM+ upon last testing)
* Use of medications that may cause increase in serum aminotransferase levels (e.g. HMG co-A reductase inhibitors, anti-epileptics, etc.) within 30 days prior to enrollment
* Any chronic or active inflammatory disease that may potentially be associated with higher inflammatory markers (examples include, but not limited to: tuberculosis, inflammatory bowel disease, pneumonia, autoimmune disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are newly diagnosed with Hepatitis C
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Determine the association between CB-CAP levels and liver fibrosis | 5 years

SECONDARY OUTCOMES:
Determine the effect of HCV treatment upon CB-CAP levels | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Butt, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States